CLINICAL TRIAL: NCT06825442
Title: AAGL 2021 Classification System And Risk Of Surgical Complications In Women Undergoing Surgery For Endometriosis
Brief Title: AAGL 2021 Classification and Surgical Complications in Women With Endometriosis
Status: Not yet recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: ENDOCHIR
Record Dates: First submitted 2025-01-10; First posted 2025-02-13 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2024-11

CONDITIONS: Endometriosis
Keywords: endometriosis; surgery; surgical complications; AAGL Classification 2021
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Several classifications exist to describe peri-operative complications including the Clavien-Dindo classification which is easily applicable to laparoscopic removal of endometriosis in all stages and is widely recommended for the evaluation of outcomes of endometriosis surgery. The most widely used staging system is the one reviewed by the American Society of Reproductive Medicine (rASRM) which, however, does not study DIE. In contrast, the ENZIAN score studies the anterior, posterior and lateral compartment of the pelvis and provides more reliable information on the extent of lesions. On the other hand, the rASRM and ENZIAN classification systems expressing the disease burden only indirectly correlate with the risk of postoperative complications and are not good predictors of post-surgical complications [19].

There are no studies in the literature evaluating the association of these complications with aspects such as the technical difficulty of surgical removal of endometriosis in relation to the extent of the disease.

The study of perioperative complications is essential in endometriosis surgery, so having a classification system capable of predicting complications on the basis of surgical complexity could guide clinical practice and post-operative management of patients with DIE.

This study could provide useful elements not only to improve the post-operative outcome of the operated patients, but also to identify preoperatively those pictures of DIE for which the surgeon will have to pay more attention because they have a higher risk of perioperative adverse events.

DETAILED DESCRIPTION:
Endometriosis is a benign chronic inflammatory disease associated with pelvic pain and subfertility, characterised by endometrial tissue located outside the uterus. Deep endometriosis (deep infiltrating endometriosis, DIE), the most severe form of endometriosis, can be defined as the involvement of anatomical organs and tissues by endometriotic lesions, regardless of the depth of infiltration.

The first therapeutic approach for deep endometriosis is hormone therapy; surgery should be limited to patients who have not responded or have intolerance to medical therapy, infertile patients with failed attempts at assisted reproductive technologies, or patients with critical ureteral or intestinal stenosis. Although complete removal of the disease has proven effective in reducing pain and improving fertility results, surgical complications can occur in 3% to 22% of cases and can drastically reduce patients' quality of life.

Several intraoperative staging systems for endometriosis have been proposed. However, there is a lack of a scoring system that accurately describes the disease burden. Recently, the American Association of Gynecologic Laparoscopists (AAGL) has developed and validated an anatomy-based grading system for intraoperative scoring of surgical complexity, using a qualitative index scale as a reference that identifies a score and also allows the assignment of a surgical complexity stage.

There are no studies in the literature evaluating the association of these complications with aspects such as the technical difficulty of surgical removal of endometriosis in relation to the extent of the disease. The study of perioperative complications is imperative in endometriosis surgery, so having a classification system capable of predicting complications on the basis of surgical complexity could guide clinical practice and post-operative management of patients with DIE.

This study could provide useful elements not only to improve the post-operative outcome of operated patients but also to identify preoperatively those DIE pictures for which the surgeon will have to pay more attention because they have a higher risk of perioperative adverse events.

ELIGIBILITY:
Inclusion Criteria:

* 18 years to 55 years;
* Pelvic ultrasound and/or radiological (MRI/ CT scan with rectal insufflation) diagnosis of endometriosis and surgery;
* At least 90 days of follow-up after surgery;
* Acquisition of informed consent for participation in the study and processing of data

Exclusion Criteria:

* Gynaecological oncology;
* Incomplete resection of macroscopic endometriotic lesions

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women of childbearing age with endometriosis undergoing complete laparoscopic removal of endometriotic lesions between January 2018 and December 2023 consecutively
Sampling Method: Non-Probability Sample
Enrollment: 198 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2025-03-02 (Estimated); Study Completion 2025-05-02 (Estimated)

PRIMARY OUTCOMES:
Association between AAGL staging and the occurrence of peri-operative complications | within 90 days from surgery
  Occurrence of (one or more) peri-operative complications

SECONDARY OUTCOMES:
Association between the AAGL score, ENZIAN classification, r-ASRM stage and the occurrence of peri-operative complications | within 90 days from surgery
  Occurrence of (one or more) peri-operative complications
Occurrence of peri-operative complications in patients undergoing surgery for DIE compared to patients undergoing surgery for DIE with hysterectomy | within 90 days from surgery
  Occurrence of (one or more) peri-operative complications
Occurrence of peri-operative complications in patients who underwent preoperative medical therapy compared to patients who did not | within 90 days from surgery
  Occurrence of (one or more) peri-operative complications
Occurrence of peri-operative complications in patients who underwent peri-operative medical therapy compared to patients who discontinued medical therapy close to surgery | within 90 days from surgery
  Occurrence of (one or more) peri-operative complications
Occurrence of clinical/radiological recurrence of disease at 24 months in patients who underwent peri-operative medical therapy compared to patients who discontinued medical therapy close to surgery | 24 months after surgery
  Onset of disease recurrence
Association between AAGL score and achievement of pregnancy (spontaneous and non-spontaneous) | At 3, 6, 9, 12, 24 and 36 months after surgery
  Onset of pregnancy

CONTACTS AND LOCATIONS:
Overall Officials: Diego Raimondo, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Italy